CLINICAL TRIAL: NCT00161629
Title: A Phase 1 Dose-Escalating, Double-Blind, Placebo-Controlled, Multicenter, Safety and Feasibility Study of Recombinant Human Bone Morphogenetic Protein-2 (rhBMP-2)/Calcium Phosphate Matrix (CPM) as an Adjuvant Therapy for Closed Distal Radius Fractures
Brief Title: Study Evaluating rhBMP-2/CPM in Closed Distal Radius Fractures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3100N7-114
Record Dates: First submitted 2005-09-01; First posted 2005-09-12 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Radius Fractures
Keywords: Distal Radius Fractures
MeSH Terms: conditions — Radius Fractures; Wrist Fractures

INTERVENTIONS:
Drug: rhBMP-2/CPM

SUMMARY:
To evaluate the safety of rhBMP-2/CPM administered to subjects presenting with closed distal radius fractures. The key safety variables comprising this assessment are: 1) incidence of delayed union; 2) median time to fracture union (assessed by the investigators); 3) incidence of local neurovascular events (those involving the region under study [RUS]); and 4) rate of fracture displacement. The primary objective will be met if these outcomes in the active and placebo treatment groups are at least comparable to those of the SOC control group.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 to 80 years of age; alert and oriented to person, place, and time.
* Acute, closed distal radius fractures (within 4 cm of the tip of the radial styloid process), classified according to AO/ASIF as either A2 or A3 (extra-articular) or C1 or C2 (intra-articular) fractures.
* Closed fracture reduction and definitive fracture fixation performed within 7 days after injury by means of external skeletal and/or percutaneous pin fixation. Note: fractures that are initially treated by closed reduction and casting, then converted to external or percutaneous pin fixation for definitive fracture fixation within 7 days after injury are eligible for the study.

Other inclusion applies.

Exclusion Criteria:

* Other fractures of the ipsilateral upper extremity (except for ulnar styloid fractures) or the contralateral upper extremity (except for previously healed fractures without residual functional deficit).
* Fracture fixation by other means (eg, plate and screw fixation).
* Planned treatment for the fracture includes any procedure to promote fracture healing (eg, open reduction internal fixation, bone grafting, non-invasive modalities such as ultrasound, electrical stimulation, etc). Note: After 12 weeks have elapsed since administration of the treatment assignment, unanticipated procedures to promote fracture healing are permitted as clinically indicated.

Other exclusion applies.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Determine the safety of administering rhBMP-2/CPM to subjects with distal radius fractures that require surgical fixation.

SECONDARY OUTCOMES:
Feasibility of the test article injection procedure and localization of the test article relative to the distal radius fracture site.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Finland, MedInfoNord@wyeth.com
Locations (5):
- Finland (3):
  - Kuopio
  - Oulu
  - Turku
- France (2):
  - Créteil
  - Paris